CLINICAL TRIAL: NCT00002943
Title: High Dose Carboplatin, Etoposide, Cyclophosphamide and Autologous Bone Marrow Transplantation for Relapsed and Refractory Germ Cell Cancer: A Phase II Pilot Study
Brief Title: Carboplatin, Etoposide, Cyclophosphamide, and Autologous Bone Marrow Transplantation in Patients With Relapsed or Refractory Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000065392; CCCWFU-95193; NCI-G97-1146
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Extragonadal Germ Cell Tumor; Ovarian Cancer; Testicular Germ Cell Tumor; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage III malignant testicular germ cell tumor; recurrent malignant testicular germ cell tumor; unspecified adult solid tumor, protocol specific; stage III ovarian germ cell tumor; stage IV ovarian germ cell tumor; recurrent ovarian germ cell tumor; extragonadal germ cell tumor
MeSH Terms: conditions — Ovarian Neoplasms; Testicular Germ Cell Tumor; Testicular Neoplasms | interventions — Carboplatin; Cyclophosphamide; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: carboplatin
Drug: cyclophosphamide
Drug: etoposide
Procedure: autologous bone marrow transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining chemotherapy with autologous bone marrow transplantation may help the body kill more tumor cells.

PURPOSE: Phase II trial to study the effects of high doses of carboplatin, etoposide, and cyclophosphamide followed by autologous bone marrow transplantation in patients with relapsed or refractory germ cell cancer and other chemotherapy-sensitive solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

* Investigate the response rate, duration of response, survival, time to marrow reconstitution, and toxicity of two successive cycles of high dose carboplatin, etoposide, and cyclophosphamide chemotherapy and ABMT in patients with relapsed and refractory germ cell cancer or other chemotherapy-sensitive solid tumors.
* Further define the pretransplant characteristics of patients and their disease that might influence the outcome of this therapy.

OUTLINE: Patients receive carboplatin and etoposide for 5 days and cyclophosphamide for 2 days prior to ABMT.

At day 60 following ABMT, if the patient has a complete response (CR) or partial response (PR) and nonhematologic toxicity is no greater than grade 2, a second ABMT course is given when hematologic parameters and other criteria are acceptable. If there is no CR or PR and/or nonhematologic toxicity exceeds grade 2, a second ABMT is not given.

After ABMT patients are followed until disease progression or death.

PROJECTED ACCRUAL: Ten patients will be accrued for this pilot study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed, measurable germ cell cancer relapsed or refractory after frontline therapy with cisplatin and etoposide-containing chemotherapy
* Other chemotherapy-sensitive solid tumors eligible (as of 06/11/97)
* Possibility of residual mass representing benign teratoma must be excluded
* Elevated serum tumor markers only are acceptable if possibilities of false-positive serum tumor markers or sanctuary disease have been excluded
* Also eligible after two to four cycles of conventional dose salvage chemotherapy, regardless of response
* No CNS or bone marrow involvement

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Karnofsky 60-100%

Life expectancy:

* Greater than 2 months

Hematopoietic:

* Platelet count at least 100,000/mm3
* Neutrophil count at least 1,500/mm3

Hepatic:

* Bilirubin, alkaline phosphatase, SGOT, and SGPT less than 3 times upper limit of normal, unless due to disease

Renal:

* Creatinine less than 1.5 times upper limit of normal
* Creatinine clearance at least 60 ml/min

Cardiovascular:

* Ventricular ejection fraction at least 45%
* No uncontrolled or severe cardiovascular disease including recent myocardial infarction, congestive heart failure, angina, life-threatening arrhythmia, or hypertension

Pulmonary:

* DLCO and spirometry greater than 50% of predicted

Other:

* Not HIV positive
* No active peptic ulcer
* No uncontrolled diabetes mellitus
* No active infection
* No previous or concomitant malignancy other than curatively treated basal or squamous cell carcinoma of the skin
* Not HBsAG positive

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior high-dose carboplatin, etoposide, or cyclophosphamide

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 1993-02; Primary Completion 2003-10 (Actual); Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
To investigate the response rate High Dose Carboplatin, Etoposide, Cyclophosphamide and Autologous Transplantation | 45 days

SECONDARY OUTCOMES:
evaluate toxicity of High Dose Carboplatin, Etoposide, Cyclophosphamide and Autologous Transplantation | 45 days

CONTACTS AND LOCATIONS:
Overall Officials: David D. Hurd, MD, Study Chair — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center at Wake Forest University, Winston-Salem, North Carolina, United States